CLINICAL TRIAL: NCT00654225
Title: A 6-Week, Randomized,Open-Label, Comparative Study to Evaluate the Efficacy and Safety of Rosuvastatin and Atorvastatin in the Treatment of Hypercholesterolaemia in South Asian Subjects.
Brief Title: Treatment of Hypercholesterolaemia in South Asian Subjects (IRIS)
Acronym: IRIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522US/0006; D3560L00026
Record Dates: First submitted 2008-03-26; First posted 2008-04-07 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia; Dyslipidaemia
Keywords: Cholesterol; low density lipoproteins; dyslipidaemia; Rosuvastatin; Crestor; Atorvastatin; Lipitor; South Asian
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Rosuvastatin Calcium; Atorvastatin

ARMS (2):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effect of 6 weeks of treatment with Rosuvastatin with 6 weeks of treatment with Atorvastatin in South Asian subjects with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Fasting low density lipoprotein & triglyceride levels as defined by the protocol.
* Self described South Asian race
* Subjects with coronary heart disease or at high risk of coronary heart disease.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Blood lipid levels above the limits defined in the protocol.
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2340 (Estimated)
Dates: Start 2002-10; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Low density lipoproteins cholesterol levels | 6 weeks

SECONDARY OUTCOMES:
Safety: adverse events & abnormal laboratory markers | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prashkrah Deedwania, Principal Investigator — Institute for Medical consultation, USA; Russell Esterline, Study Director — AstraZeneca